CLINICAL TRIAL: NCT05263518
Title: Influence of Different Toric Intraocular Lenses on IOL-capsular Complex After Cataract Surgery
Brief Title: Influence of Different Toric Intraocular Lenses on IOL-capsular Complex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TORIC stability
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Corneal Astigmatism; Cataract
Keywords: Various Types of toric IOLs
MeSH Terms: conditions — Astigmatism; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AcrySof IQ toric IOL (Experimental): patients who had cataract surgery with AcrySof IQ toric IOL implantation. The patients diagnosed age related cataract The patients' ages are over 50.
  Interventions: Procedure: Cataract surgery with AcrySof IQ IOL implantation.
- TECNIS toric IOL (Experimental): patients who had cataract surgery with TECNIS toric IOL implantation. The patients are diagnosed age related cataract. The patients' ages are over 50.
  Interventions: Procedure: Cataract surgery with TECNIS toric IOL implantation.

INTERVENTIONS:
Procedure: Cataract surgery with AcrySof IQ IOL implantation. — Patients in this study will receive cataract surgery with AcrySof IQ IOL implantation.
  Arms: AcrySof IQ toric IOL
Procedure: Cataract surgery with TECNIS toric IOL implantation. — Patients in this study will receive cataract surgery with TECNIS toric IOL implantation.
  Arms: TECNIS toric IOL

SUMMARY:
Corneal astigmatism is refractive error that impairs uncorrected visual acuity. When patients undergo cataract surgery, implantation of toric IOL is deemed the most effective choice for correcting corneal astigmatism and reducing postoperative spectacle dependence. The IOL-capsular complex is formed after cataract surgery and intraocular lens (IOL) implantation. Early postoperative mechanical wrapping of the anterior and posterior capsules plays a significant role in preventing IOL decentration and tilt, as well as formation of the IOL-capsular complex which reduces the incidence of posterior cataract opacity. IOL decentration ≥ 0.4 mm or/and IOL tilt ≥7degree were considered clinically significant because of poor post-surgery visual quality especially for optical sophisticated IOLs such as toric IOLs. IOL instability could decrease the curative effect of toric IOL. There are numerous types of toric IOLs; however, AcrySof IQ and TECNIS toric IOL are most frequently used in the Ophthalmology Hospital of Wenzhou Medical University. AcrySof IQ IOL has some differences compared with TECNIS toric IOL. IQ has a modified L haptic design while TECNIS® toric IOL has a modified C haptic design. AcrySof IQ IOL has a discontinuous 360˚ posterior square edge while TECNIS toric IOL has a continuous 360˚ posterior square edge. The AcrySof IQ IOL cylinder power models include 1.00, 1.50, 2.25, 3.00, 3.75, 4.50, 5.25 and 6.00 D. The Tecnis IOL cylinder power models include 1.00, 1.50, 2.25, 3.00 and 4.00 D. Previous study pointed that patients with cataracts with corneal astigmatism achieved comparable improvement in visual acuity, astigmatism correction, CS（sensitive contrast）, rotational stability and satisfaction, following AcrySof and TECNIS toric IOL implantation. However，some other studies found that the Acrysof toric IOL showed significantly greater rotational stability than the Tecnis toric IOL and the rate of surgical IOL repositioning was higher in eyes implanted with TECNIS than with AcrySof toric IOLs for astigmatic correction. Currently, there is no literature guidance to compare the results of cataract surgery combined various types of toric IOLs implantation in patients using CASIA2. The novel anterior segment optical coherence tomography (AS-OCT) device, CASIA2 can accurately evaluate the IOL capsule bending and the lens position after cataract surgery. Also, CASIA2 can be used to documented the dynamic changes of IOL-capsular complex after surgery.

DETAILED DESCRIPTION:
Corneal astigmatism is refractive error that impairs uncorrected visual acuity. When patients undergo cataract surgery, implantation of toric IOL is deemed the most effective choice for correcting corneal astigmatism and reducing postoperative spectacle dependence. The IOL-capsular complex is formed after cataract surgery and intraocular lens (IOL) implantation. Early postoperative mechanical wrapping of the anterior and posterior capsules plays a significant role in preventing IOL decentration and tilt, as well as formation of the IOL-capsular complex which reduces the incidence of posterior cataract opacity.

Although up to 2-3 degree tilt and a 0.2-0.3 mm decentration are common and clinically unnoticed for any design of IOL, larger extent of tilt and decentration has a negative impact on the optical performance. IOL decentration ≥ 0.4 mm or/and IOL tilt ≥7degree were considered clinically significant because of poor post-surgery visual quality especially for optical sophisticated IOLs such as toric IOLs. IOL instability could decrease the curative effect of toric IOL. There are numerous types of toric IOLs; however, AcrySof IQ and TECNIS toric IOL are most frequently used in the Ophthalmology Hospital of Wenzhou Medical University. AcrySof IQ IOL has some differences compared with TECNIS toric IOL. IQ has a modified L haptic design while TECNIS® toric IOL has a modified C haptic design. AcrySof IQ IOL has a discontinuous 360˚ posterior square edge while TECNIS toric IOL has a continuous 360˚ posterior square edge. The AcrySof IQ IOL cylinder power models include 1.00, 1.50, 2.25, 3.00, 3.75, 4.50, 5.25 and 6.00 D. The Tecnis IOL cylinder power models include 1.00, 1.50, 2.25, 3.00 and 4.00 D. Previous study pointed that patients with cataracts with corneal astigmatism achieved comparable improvement in visual acuity, astigmatism correction, CS（sensitive contrast）, rotational stability and satisfaction, following AcrySof and TECNIS toric IOL implantation. However，some other studies found that the Acrysof toric IOL showed significantly greater rotational stability than the Tecnis toric IOL and the rate of surgical IOL repositioning was higher in eyes implanted with TECNIS than with AcrySof toric IOLs for astigmatic correction. Currently, there is no literature guidance to compare the results of cataract surgery combined various types of toric IOLs implantation in patients using CASIA2. The novel anterior segment optical coherence tomography (AS-OCT) device, CASIA2 can accurately evaluate the IOL capsule bending and the lens position after cataract surgery. Also, CASIA2 can be used to documented the dynamic changes of IOL-capsular complex after surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patients are diagnosed age related cataract or complicated with corneal astigmatism
* The patients' age over 50 years old
* The patients plan to receive cataract surgery in Eye hospital of Wenzhou Medical University
* The dilated pupils are over 7mm
* Patients are willing and able to complete the follow-ups.

Exclusion Criteria:

* Patients with other type of cataract
* Patients have complications in the surgery and after surgery
* Patients have other severe diseases of eyes

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The position of IOL | The 1st day after surgery
  Evaluation of the position of IOL through tilt, decentration，rotation and the process of capsule bending using CAISA2（The novel anterior segment optical coherence tomography (AS-OCT) device）
The position of IOL | The 1st week after surgery
  Evaluation of the position of IOL through tilt, decentration，rotation and the process of capsule bending using CAISA2（The novel anterior segment optical coherence tomography (AS-OCT) device）
The position of IOL | The 1st month after surgery
  Evaluation of the position of IOL through tilt, decentration，rotation and the process of capsule bending using CAISA2（The novel anterior segment optical coherence tomography (AS-OCT) device）
The position of IOL | The 3rd month after surgery
  Evaluation of the position of IOL through tilt, decentration，rotation and the process of capsule bending using CAISA2（The novel anterior segment optical coherence tomography (AS-OCT) device）

CONTACTS AND LOCATIONS:
Overall Officials: Yune Zhao, Study Director — Ophthalmology and Optometry Hospital

REFERENCES:
- [Derived] Wang Y, Lou X, Qian S, Li Y, Wu X, Li S, Wang Y, Zhao Y, Chang P. Comparison of the effect of capsular bend on the rotational stability between 2 toric intraocular lenses. J Cataract Refract Surg. 2024 Mar 1;50(3):283-288. doi: 10.1097/j.jcrs.0000000000001373. PMID 38085243